CLINICAL TRIAL: NCT01068938
Title: Detection of Visual Field Defects and Scotoma Progression in Glaucomatous Optic Neuropathy, Using Short-term Intervals With Automated Scotoma-oriented Perimetry (SCOPE) and the Fast Thresholding Strategy GATE (German Adaptive Threshold Estimation)
Brief Title: Comparison of Visual Fields: Humphrey Field Analyzer (HFA) SITA Strategy, SCOPE (GATE Strategy) and Humphrey MATRIX Perimeter
Acronym: X-SCOPE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ulrich Schiefer, Prof. Dr. med., University Hospital Tuebingen
Other Study IDs: X-SCOPE; 116MIR08023 (Other Grant/Funding Number: Pfizer); 428/2008BO1 (Other: Ethics Committee University Hospital Tübingen)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Glaucoma
Keywords: visual field; perimetry; glaucoma progression; grid; POAG and glaucoma suspects with prostaglandin monotherapy
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- open angle glaucoma, glaucoma suspects: risk of progression, Latanoprost monotherapy
  Interventions: Device: three different perimeters: HFA, Octopus, MATRIX

INTERVENTIONS:
Device: three different perimeters: HFA, Octopus, MATRIX — visual fields

SUMMARY:
The purpose of this study is to compare three perimetric techniques regarding progression of the visual field.

ELIGIBILITY:
Inclusion Criteria:

* max. ± 8 dpt sph, max. ± 3 dpt cyl
* distant visual acuity > 10/20
* isocoria, pupil diameter > 3 mm
* at least one risk of progression: optic disc (splinter) hemorrhage / cup to disc ratio (CDR) > 0.7 / inter-eye asymmetry of CDR >0.2 / notching of the optic disc /retinal nerve fibre layer (RNFL) defects / intraocular pressure( IOP) >22 mmHg / central corneal thickness < 520 µm / advanced visual field defect stage Aulhorn III / elder than 70 years

Exclusion Criteria:

* pregnancy, nursing
* diabetic retinopathy
* asthma
* HIV+ or AIDS
* history of epilepsy or significant psychiatric disease
* medications known to effect visual field sensitivity
* infections (e.g. keratitis, conjunctivitis, uveitis)
* severe dry eyes
* miotic drug
* amblyopia
* squint
* nystagmus
* albinism
* any ocular pathology, in either eye, that may interfere with the ability to obtain visual fields,disc imaging or accurate IOP readings
* keratoconus
* intraocular surgery (except for uncomplicated cataract surgery) performed < 3 month prior to screening
* history or signs of any visual pathway affection other than glaucoma
* allergies with regard to topic glaucoma medication
* history or presence of macular disease and / or macular edema
* ocular trauma
* medications known to affect visual field sensitivity

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University Eye Hospital
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
glaucoma progression | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, MD, Principal Investigator — Centre for Ophthalmology, Institute for Ophthalmic Research
Locations (1):
- Centre for Ophthalmology, Institute for Ophthalmic Research, Tübingen, Germany

REFERENCES:
- [Background] Schiefer U, Pascual JP, Edmunds B, Feudner E, Hoffmann EM, Johnson CA, Lagreze WA, Pfeiffer N, Sample PA, Staubach F, Weleber RG, Vonthein R, Krapp E, Paetzold J. Comparison of the new perimetric GATE strategy with conventional full-threshold and SITA standard strategies. Invest Ophthalmol Vis Sci. 2009 Jan;50(1):488-94. doi: 10.1167/iovs.08-2229. Epub 2008 Dec 5. PMID 19060285
- See also: Publication — http://iovs.arvojournals.org/article.aspx?articleid=2125766